CLINICAL TRIAL: NCT00960479
Title: A Relative Bioavailability Study of Ribavirin (Geneva Pharmaceutical Technology Corporation, N.J., U.S.A.) 200 Capsules and Rebetol (Schering Corporation, N.J., U.S.A.) 200 mg Capsules in Females Under Fasting Conditions.
Brief Title: Relative Bioavailability Study of Ribavirin 200 Capsules and Rebetol 200 mg Capsules in Females Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P1BH00001
Record Dates: First submitted 2009-08-13; First posted 2009-08-17 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-08

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin

ARMS (2):
- 1 (Experimental): Ribavirin 200 mg Oral Capsule (Geneva Pharmaceutical, U.S.A.)
  Interventions: Drug: Ribavirin 200 mg Oral Capsule (Geneva Pharmaceutical, U.S.A.)
- 2 (Active Comparator): Rebetol 200 mg Oral Capsule (Schering Corporation, U.S.A.)
  Interventions: Drug: Rebetol 200 mg Oral Capsule (Schering Corporation, U.S.A.)

INTERVENTIONS:
Drug: Ribavirin 200 mg Oral Capsule (Geneva Pharmaceutical, U.S.A.)
  Arms: 1
Drug: Rebetol 200 mg Oral Capsule (Schering Corporation, U.S.A.)
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the relative bioavailability of Ribavirin 200 capsules and Rebetol 200 mg capsules in females under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2001-01; Primary Completion 2001-02 (Actual); Study Completion 2001-02 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Piyush Patel, M.D., Principal Investigator — Allied Clinical Research